CLINICAL TRIAL: NCT06997484
Title: A Randomized, Double-blind, Placebo-controlled, Sequential Parallel Group, Single and Multiple Ascending Dose (SAD/MAD) Study in Healthy Subjects to Evaluate the Safety, Tolerability, Pharmacokinetics of HL-400 Following Oral Administration
Brief Title: First-in-Human Single and Multiple Dose of HL-400
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Highlightll Pharmaceutical (USA) LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HL-400-101
Record Dates: First submitted 2025-05-13; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HL-400 (Active Comparator): Part 1:Experimental: Single oral dose of HL-400, Single ascending doses, sequential assignment group design; Part 2: Experimental: Multiple oral doses of HL-400, Multiple ascending doses, once a day (QD) for 14 days, sequential assignment group design; Part 3: Experimental: Multiple oral doses of HL-400, QD for 5 days.
  Interventions: Drug: HL-400
- Placebo (Placebo Comparator): Part 1: Placebo comparator: Single oral dose of placebo, single doses, matching placebo; Part 2: Placebo comparator: Multiple oral doses of placebo, multiple ascending doses, QD for 14 days, matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HL-400 — Part 1:Experimental: Single oral dose of HL-400, Single ascending doses, sequential assignment group design; Part 2: Experimental: Multiple oral doses of HL-400, Multiple ascending doses, QD for 14 days, sequential assignment group design; Part 3: Experimental: Multiple oral doses of HL-400, QD for 5 days.
  Arms: HL-400
Drug: Placebo — Part 1: Placebo comparator: Single oral dose of placebo, single doses, matching placebo; Part 2: Placebo comparator: Multiple oral doses of placebo, multiple ascending doses, QD for 14 days, matching placebo.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, dose-escalation study in healthy subjects to evaluate the safety, tolerability, pharmacokinetics of HL-400 (a NLRP3 inhibitor) following oral single and multiple ascending dose administration.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, dose-escalation study in healthy subjects to evaluate the safety, tolerability, pharmacokinetics of HL-400 following oral single and multiple ascending dose administration.This study will consist of 3 parts, which are Part 1 (Single Ascending Dose), Part 2 (Multiple Ascending Dose) and Part3 (cerebrospinal fluid (CSF) Exposure).

Safety, pharmacokinetic parameters and relevant biomarkers will be assessed in the study.

ELIGIBILITY:
Inclusion Criteria:

* Are capable of giving written informed consent and complying with study procedures, schedule, requirements, and restrictions.
* Are between the ages of 18 and 65 years, inclusive, at screening.
* Female subjects have a negative serum hCG pregnancy test result at screening andDay （-1）, agree to refrain from ova donation for at least 3 months after the last dose, and willingness to comply with protocol-specified contraceptive methods.
* Male subjects with female partners of reproductive potential must agree to practice abstinence or to use a condom (male subject) plus an additional barrier method (female partner) of contraception for the duration of the study and for at least 3 months after last dosing; must also agree to refrain from sperm donation for at least 3 months after the last dose.
* Considered healthy by the Investigator, based on subject's reported medical history, full physical examination, clinical laboratory tests, 12-lead ECG, and vital signs.
* Non-smoker for at least 6 months prior to screening.
* Body mass index (BMI) of 18.0 to 32.0 kg/m2 inclusive and body weight not less than 50 kg.

Exclusion Criteria:

* Clinically significant history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders, or drug hypersensitivity as determined by the Investigator.
* Pregnant (as determined by pregnancy test result) or breastfeeding women.
* History of chronic diarrhea, malabsorption, unexplained weight loss, food allergies or intolerance.
* Positive blood screen for human immunodeficiency virus (HIV 1/2), hepatitis B surface antigen (HBsAg), or hepatitis C antibody.
* A positive screen for alcohol or drugs of abuse at screening or Day -1.
* An unwillingness or inability to comply with food and beverage restrictions during study participation.
* Volunteers who have participated in any investigational drug or device study within past 3 months prior to dosing.
* Any condition or finding that in the Investigators opinion would put the subject or study conduct at risk if the subject were to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Number and percentage of participants with adverse events (AEs) | From the time of taking first dose of study drug to 7 days after the last dose.
  To evaluate the safety and tolerability of HL-400 following oral single and multiple ascending dose administration.
Number and percentage of adverse events (AEs) according to severity | From the time of taking first dose of study drug to 7 days after the last dose.
  To evaluate the safety and tolerability of HL-400 following oral single and multiple ascending dose administration.
Change in 12-lead electrocardiogram (ECG) parameters (PR Interval, QRS Complex, QT Interval, QTC Interval) from baseline | From baseline to 7 days after the last dose.
  To evaluate the safety and tolerability of HL-400 following oral single and multiple ascending dose administration.
Single Ascending Dose (SAD) Cohorts: Maximum observed plasma concentration (Cmax) of HL-400 | From 0.5 hour to 72 hours post-dose.
  To characterize the PK in the plasma of HL-400 following oral single dose administration.
Single Ascending Dose (SAD) Cohorts: Time to reach maximum observed plasma concentration (Tmax) of HL-400 | From 0.5 hour to 72 hours post-dose.
  To characterize the PK in the plasma of HL-400 following oral single dose administration.
Single Ascending Dose (SAD) Cohorts: Plasma decay half-life (t1/2) of HL-400 | From 0.5 hour to 72 hours post-dose.
  To characterize the PK in the plasma of HL-400 following oral single dose administration.
Single Ascending Dose (SAD) Cohorts: Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUCinf) of HL-400 | From 0.5 hour to 72 hours post-dose.
  To characterize the PK in the plasma of HL-400 following oral single dose administration.
Multiple Ascending Dose (MAD) Cohorts: Maximum observed plasma concentration (Cmax) of HL-400 | From Day 1 pre-dose to 72 hours after the last dose.
  To characterize the PK in the plasma of HL-400 following oral multiple ascending dose administration.
Multiple Ascending Dose (MAD) Cohorts: Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUCinf) of HL-400 | From Day 1 pre-dose to 72 hours after the last dose.
  To characterize the PK in the plasma of HL-400 following oral multiple ascending dose administration.

SECONDARY OUTCOMES:
1.The cerebrospinal fluid (CSF) cohort: Maximum observed concentration (Cmax) of HL-400 in the CSF | From Day 1 pre-dose to 24 hours after the last dose
  To characterize the PK in the CSF of HL-400 following oral multiple dose administration.
The cerebrospinal fluid (CSF) cohort: Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUCinf) of HL-400 in the CSF | From Day 1 pre-dose to 24 hours after the last dose
  To characterize the PK in the CSF of HL-400 following oral multiple dose administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaron CPC, Inc., Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No